# AcelRx Pharmaceuticals, Inc.

#### PROTOCOL No. IAP312

A Multicenter, Open-Label Trial to Evaluate the Overall Performance of the Zalviso System (sufentanil sublingual tablet system) 15 mcg

Statistical Analysis Plan for Final Data Analysis

(Final Version, 6/10/2017)

| Prepared by: | | |
|---|---|---|
| | Yu-Kun Chiang, PhD<br>Statistical Consultant to AcelRx | Date |
| AcelRx:<br>Approved by: | | |
| | Pamela Palmer, M.D., Ph.D. Chief Medical Officer | Date |

# **TABLE OF CONTENTS**

| | | Page |
|---|---|---|
| 1 | Introduction | 1 |
| 2 | Statistical Methods | 1 |
| 2.1 | Determination of Sample Size | 1 |
| 2.2 | Data Processing and Management | 1 |
| 2.3 | Performance of Statistical Data Analysis | 1 |
| 2.4 | Protocol Deviations and Special Cases | 2 |
| 2.5 | Test of Hypothesis and Significance Levels | 2 |
| 2.6 | Randomization and Blinding of Treatment Assignment | 2 |
| 2.7 | Patient Enrollment and Disposition | 2 |
| 2.8 | Premature Termination from the Study | 2 |
| 2.9 | Baseline Comparability | 2 |
| 2.10 | Analysis of Efficacy Data | 2 |
| 2.10.1 | Efficacy Variables | 2 |
| 2.10.2 | Analysis Population and Handling of Dropouts | 3 |
| 2.10.3 | Definition of Baseline Measurements | 4 |
| 2.10.4 | Methods for the Analysis of Device Dispense Failure Rate | 4 |
| 2.10.5 | Pooling of Investigators | 5 |
| 2.10.6 | Methods for the Analysis of Categorical Efficacy Variables | 5 |
| 2.10.7 | Methods for the Analysis of Continuous Efficacy Variables | 5 |
| 2.11 | Analysis of Safety Data | 6 |
| 2.11.1 | Extent of Exposure to Study Drug | 6 |
| 2.11.2 | Adverse Events | 6 |
| 2.11.3 | Death Reports and Serious Adverse Events | 6 |
| 2.11.4 | Adverse Events Causing Premature Discontinuation of Study Drug | 6 |
| 2.11.5 | Summary of Adverse Events by Severity and Relationship to Study Drug . | 7 |
| 2.11.6 | Subgroup Summary of Adverse Events | 7 |
| 2.11.7 | Pregnancy Test Results | 7 |
| 2.11.8 | Vital Signs | |
| 2.11.9 | Physical Examination Data | 7 |
| 2.11.10 | 0 Concomitant Medications | 7 |
| 2.12 | Handling of Partial Dates and Partial Times | 8 |
| 2.13 | The Presentation of Data Listings | 8 |
| 2.14 | Computer Software | 9 |
| | References | 9 |

i

# Protocol No. IAP312: FINAL REPORT Statistical Analysis Plan

| Table A-1 | Evaluation Time Points with Evaluation Windows Used for the Summary of Global Assessment Data by Evaluation Time Point | |
|---|---|---|
| Table A-2 | Scheduled Evaluation Time Points with Evaluation Windows Used for the Summary of Pain Assessment Data, Blood Pressures, and Heart Rates by Evaluation Time Point | .11 |
| Table A-3 | Scheduled Evaluation Time Points with Evaluation Windows Used for the Summary of Respiratory Rates and Oxygen Saturation Data by Evaluation Time Point | .13 |

#### 1 Introduction

This is a multicenter, open-label, single treatment clinical study designed to evaluate the overall functionality of the Zalviso System (sufentanil sublingual tablet system) 15 mcg for the treatment of acute moderate-to-severe postoperative pain.

The study was designed to demonstrate that the device dispense failure rate is non-inferior to a target of 2%. This is based on the criteria that the upper limit of a 90% confidence interval (CI) of the device dispense failure rate is not worse than 5%.

The statistical issues regarding the conduct and analysis of this study are described briefly in the following sections.

#### 2 Statistical Methods

#### 2.1 Determination of Sample Size

A sample size of approximately 330 patients is planned for this study in order to have at least 315 patients receive study drug and have available efficacy data for data analysis.

A sample size of 315 patients will have 90% power to demonstrate that the device dispense failure rate is non-inferior to a target of 2%. This failure rate is the proportion of patients who experienced at least one of following events: (1) a system-generated error, (2) a tablet dispensed but not requested, or (3) a tablet dispensed when the Zalviso System is in lockout. All events listed above will be obtained from the Controller patient usage data.

This is based on the criteria that the upper limit of a 90% confidence interval (CI) of the device dispense failure rate is not worse than 5%. This calculation is based on the exact binomial test of one-sample proportion for a one-sided case against a 2% target proportion with a delta of 3%, and a one-sided significance level of  $\alpha$ =0.05. This sample size was generated from the SAS procedure PROC POWER for one-sample proportion. Exact power computations are based on the binomial distribution and computing formulas provided by Johnson and Kotz (1970). Assuming a 5% non-evaluable rate, a sample size of 330 patients is planned for this study.

## 2.2 Data Processing and Management

All data management activities including the Case Report Form (CRF) data entry, query generation, query resolution and data base maintenance, were performed by the Data Management Department of PRA Health Sciences.

# 2.3 Performance of Statistical Data Analysis

The statistical data analysis will be performed by Essence Sciences Inc.

## 2.4 Protocol Deviations and Special Cases

Enrolled patients who deviate from the study protocol will be listed in Appendix 16.2. Protocol deviations at entry and deviations related to the efficacy measurements during the study will be identified.

# 2.5 Test of Hypothesis and Significance Levels

Both continuous and categorical efficacy variables will be summarized descriptively. A point estimate of the device dispense failure rate and its 90% exact Clopper-Pearson confidence interval will be constructed. The statistical tests for the analysis of other efficacy variables and safety data will be performed at the  $\alpha = 0.05$  significance level. All tests will be two-sided.

## 2.6 Randomization and Blinding of the Treatment Assignment

This is an open-label single treatment study. There is no randomization of patients or blinding of treatment. Patients who meet the eligibility requirements will be enrolled into this study sequentially within each study center to receive study treatment.

# 2.7 Patient Enrollment and Disposition

Post-text Table 14.1.1 summarizes the number of patients enrolled in this study by surgery type within each investigator's site. Post-text Table 14.1.2 defines the patient population used for the efficacy and safety data analysis.

#### 2.8 Premature Termination from the Study

Patients who prematurely terminate from the study will be summarized according to the reason for termination. Each unique reason will be determined by the investigator.

Patients who prematurely terminated from the study and reasons for not entering next time period will be summarized in Post-text Tables 14.1.3 to 14.1.7.

#### 2.9 Baseline Comparability

Demographics and baseline characteristics will be summarized for all enrolled patients in Post-text Table 14.1.8. Data will be pooled for all study centers for the descriptive summary of baseline data. No formal hypothesis testing will be performed for baseline data. Similar summaries will be performed for the safety population separately in Post-text Table 14.1.9.

#### 2.10 Analysis of Efficacy Data

Sections related to the analysis of efficacy data are specified below by topic.

#### 2.10.1 Efficacy Variables

The efficacy variables and parameters are:

- (1) Proportion of patients who experienced at least one system-generated error based on the Controller data while using the Zalviso System
- (2) Proportion of patients, if any, with tablet dispensed but not requested
- (3) Proportion of patients, if any, with tablet dispensed when the Zalviso System is in lockout
- (4) Proportion of patients with misplaced tablet(s)
- (5) Number of misplaced tablets (i.e., tablet found outside the patient's mouth)
- (6) Proportion of patients who experienced either a system-generated error or a misplaced tablet (i.e. a dispense failure)
- (7) Assessment of the number of Zalviso System notifications to the nurse to retrain patient to not pull down on Controller while dosing (i.e., mitigation of Error 302)
- (8) Proportion of patients who rate the Patient Global Assessment (PGA) of method of pain control over 24, 48 and 72 hours as "good" or "excellent"
- (9) Proportion of patients who responded in each category of the PGA
- (10) Proportion of Healthcare Professionals who rate the Global Assessment (HPGA) of method of pain control over 24, 48 and 72 hours as "good" or "excellent"
- (11) Proportion of Healthcare Professionals who responded in each category of the HPGA
- (12) Proportion of patients who terminate from the study due to inadequate analgesia over the 24-hour, 48-hour and 72-hour study period
- (13) Time to terminate from the study due to inadequate analgesia
- (14) Time-weighted summed pain intensity difference (SPID) over the 24-hour study period (SPID24), over the 48-hour study period (SPID48), and over the 72-hour study period (SPID72)
- (15) SPID up to each evaluation time point
- (16) Total pain relief (TOTPAR) over the 24-hour study period (TOTPAR24), over the 48-hour study period (TOTPAR48) and over the 72-hour study period (TOTPAR72)
- (17) TOTPAR up to each evaluation time point
- (18) Pain intensity (PI) at each evaluation time point
- (19) Pain intensity difference (PID) at each evaluation time point
- (20) Pain relief (PR) at each evaluation time point
- (21) Patient Usability Questionnaire (PUQ)
- (22) Nurse Usability Questionnaire (NUQ)

- (23) Total number of study drug doses used over 24, 48, and 72-hour study period, average hourly use, and average inter-dosing interval.
- (24) Total amount of supplemental morphine utilized

# 2.10.2 Analysis Population and Handling of Dropouts

All enrolled patients are those who are enrolled and receive the study treatment. The main analysis of efficacy endpoints includes all enrolled patients.

For patients missing PI or PR data, the following methods will be applied to impute the missing data at evaluation time points for the duration of study period:

- (1) Missing data will be first imputed on a patient-by-patient basis by linear interpolation method between two observed pain scale values.
- (2) Data occurring after a patient terminated from study or did not provide any follow-up data after last available data prior to the end of study period, the pain scale values at follow-up time points post-termination up to the end of the study period will be imputed on a patient-by-patient basis as described below.

The last observation carried forward (LOCF) method will be used to impute any remaining missing data points after termination due to reasons other than adverse event up to the end of the study period. For patients who prematurely terminate from the study due to adverse event, the worst observation carried forward (WOCF) method will be used to impute the remaining missing data points up to the end of the study period. The worst PID is the smaller number between number zero and the last PID obtained prior to termination. The worst PR is number zero.

For patients who use any supplemental opioid during the study period, the last observed pain intensity prior to using each dose of supplemental opioid will be carried throughout a follow-up 1-hour time interval. Any pain intensity collected within 1 hour after the start of any supplemental opioid will be excluded from the calculation of the time-weighted SPID. This same imputation method will also be used to calculate the efficacy endpoints derived from pain assessment data.

#### 2.10.3 Definition of Baseline Measurements

Baseline measurements are those taken prior to the start of study drug administration.

#### 2.10.4 Methods for the Analysis of Device Dispense Failure Rate

For the analysis of the device dispense failure rate, a point estimate of the device dispense failure rate and its 90% exact Clopper-Pearson confidence interval will be constructed. Patients from all study centers will be pooled for the descriptive summary of these efficacy data.

Results generated from the analysis of these dichotomous efficacy endpoints derived from the device performance data and misplaced tablets will be presented in Post-text Tables 14.2.1 to 14.2.7.

#### 2.10.5 Pooling of Investigators

The data collected from all study centers will be pooled for the analysis of efficacy data.

#### 2.10.6 Methods for the Analysis of Categorical Efficacy Variables

For the analysis of the dichotomous outcome data, a point estimate and its 95% confidence interval will be constructed. Patients from all study centers will be pooled for the descriptive summary of the efficacy data.

Results generated from the analysis of these categorical efficacy variables will be presented in Post-text Tables 14.2.8 to 14.2.18.

#### 2.10.7 Methods for the Analysis of Continuous Efficacy Variables

The method used to derive the efficacy endpoint time-weighted summed pain intensity difference (SPID) over the study period is described in this section. Pain intensity will be measured using an 11-point NRS with 0 (no pain) and 10 (worst possible pain).

Patients will provide the pain intensity (PI) and pain relief (PR) measures at baseline and at each evaluation time point after the initiation of the first ondemand dose of study drug: ½ [15 min], ½ [30 min], ¾ [45 min], 1, 2, 4, 6, 8, 10, and 12 hours, then every 4 hours at 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72 hours.

The PID at each evaluation time point after the initiation of the first dose is the difference in pain intensity at the specific evaluation time point and baseline pain intensity [PID (evaluation time after the first dose) = pain intensity (baseline) – pain intensity (evaluation time after the first dose)]. The time-weighted SPID24 is the time-weighted summed PID over the 24-hour study period.

Time-weighted SPID24 =  $\sum [T(i) - T(i-1)] \times PID(i)$ ,

Where : T(0) = Time 0 (baseline), T(i) is the scheduled or unscheduled assessment time, and PID(i) is the PID score at time i for i=0 to 24 hours

Other time-weighted SPID, SPID48 and SPID72 will be derived similarly. TOTPAR over follow-up evaluation time periods (e.g., TOTPAR24, TOTPAR48, and TOTPAR72, etc.) will be derived from the PR data collected during the study using similar formula described above.

For the analysis of the continuous efficacy data, a point estimate and its 95% confidence interval will be constructed. Patients from all study centers will be pooled for the descriptive summary of the efficacy data

## 2.11 Analysis of Safety Data

The safety data collected in this study include:

- (1) Adverse events(AEs)
- (2) Pregnancy test results
- (3) Vital signs
- (4) Physical examination data
- (5) Suspected technical failures
- (6) Concomitant medications

All enrolled patients who receive at least one dose of study drug will be included in the analyses and summaries of safety data.

## 2.11.1 Extent of Exposure to Study Drug

The length of exposure to study drug will be summarized in Post-text Table 14.3.1.

#### 2.11.2 Adverse Events

Adverse events occurring while patients were on study medication during the treatment period or within 12 hours after the discontinuation of study medication will be summarized in Post-text Table 14.3.2. All incidences of AEs will be summarized in Post-text Table 14.3.3. The MedDRA® (Medical Dictionary for Regulatory Activities) V11.0 thesaurus will be used to map the AE verbatim to lowest level term (LLT), preferred term (PT) and System Organ Class (SOC) for summary purposes. Adverse event data including the AE verbatim term and the associated AE thesaurus preferred term will be provided in the patient data listings.

The most frequent AEs (e.g., those in at least 1% of all treated patients) will be summarized in Post-text Table 14.3.4.

## 2.11.3 Death Reports and Serious Adverse Events

Death that occurred during the study will be listed and discussed. Serious adverse events will be summarized in Post-text Table 14.3.5

#### 2.11.4 Adverse Events Causing Premature Discontinuation of Study Drug

Adverse events causing premature discontinuation of study drug will be summarized in Post-text Table 14.3.6.

## 2.11.5 Summary of Adverse Events by Severity and Relationship to Study Drug

Adverse events will be summarized by severity and relationship to study drug (related or not related) in Post-text Table 14.3.7. Related AEs are those AEs possibly or probably related to study drug. Adverse events will be summarized by maximum severity in Post-text Table 14.3.8 and summarized by closest relationship to the study drug in Post-text Table 14.3.9. Adverse events related to the study drug, severe adverse events, and severe adverse events related to the study drug will be summarized by treatment groups in Post-text Table 14.3.10 and 14.3.12 respectively. 3.6.

## 2.11.6 Subgroup Summary of Adverse Events

Adverse events will be summarized by age group (< 65 years and  $\geq$  65 years), sex group (male and female), race group (Caucasian and Non-Caucasian), and body mass index group (< 30 kg/m² and  $\geq$  30 kg/m²) in Post-text Table 14.3.13 and 14.3.16 respectively. A two-sided Fisher's exact test will be used for the comparison among subgroups.

## 2.11.7 Pregnancy Test Results

Pregnancy test results will be listed in the Appendix.

# 2.11.8 Vital Signs

Vital signs, including blood pressure, heart rate, respiratory rates, and oxygen saturation data, taken at baseline and follow-up time points will be summarized in Post-text Tables 14.3.17 to 14.3.21. Patients who had baseline data and at least one follow-up data will be included in this analysis. The descriptive summary statistics will be presented. A paired t-test will be used for the test of mean change from baseline to follow-up time points within each group.

The lowest oxygen saturation value will be identified for each patient. Two dichotomous variables will be defined based on this lowest observed value at two cut-off levels of 93% and 95% of oxygen saturation. These lowest oxygen saturation variables will be summarized. The results of these summaries will be presented in Post-text Table 14.3.22.

#### 2.11.9 Physical Examination Data

The physical examination data will be listed in the Appendix.

#### 2.11.10 Concomitant Medications

Concomitant medications used during the study will be summarized in Post-text Table 14.3.23. Medications discontinued before the enrollment date will be

excluded from the summary. The World Health Organization (WHO) Drug Dictionary (WHO-DD, 01DEC2015 version) will be used to map the medication name to the Anatomical Therapeutic Chemical (ATC) classification codes for summary purpose.

If a medication is mapped to more than one ATC-code, a unique ATC-code will be selected based on the condition treated. The concomitant medications will be summarized by the medication category, medication class, and medication subgroup based on the ATC-codes. The medication category will be determined by the first character of the ATC-code. The medication class will be determined by the first three characters of the ATC-code. The medication subgroup will be determined by all the characters (maximum five characters) of the ATC-code.

#### 2.12 Handling of Partial Dates and Partial Times

Complete date and time values were required for certain date fields on the CRFs (e.g., assessment date and time, dosing date and time, etc.). However, partial date values may have been acceptable for selected date fields on the CRFs (e.g., start dates of concomitant medications or adverse events prior to entry). In order to calculate the duration of events, the following assumptions were applied to estimate the complete date and time values for the partial event start date and time values:

- (1) If only the "time" value was missing, the first minute (00:01) of the day was used.
- (2) If only the "day" value was missing, the first day of the month was used.
- (3) If only the "month" value was missing, January was used.
- (4) If both "day" and "month" values were missing, January first was used.

The "year" value of the date field was required for all cases. The estimated event date/time should not be later than the available event stop date/time for a given event.

For those adverse events with partial AE stop date/time and stopped prior to the study termination, the following assumptions were applied to estimate the complete date values:

- (1) If only the "time" value was missing, the last minute (23:59) of the day was used.
- (2) If only the "day" value was missing, the last day of the month was used.
- (3) If only the "month" value was missing, December was used.
- (4) If both "day" and "month" values are missing, December 31st was used.

If the estimated AE stop date/time based on the assumptions listed above was later than the study termination date, the partial AE stop date/time was estimated from the study termination date/time.

#### 2.13 The Presentation of Data Listing

In addition to the summary Tables presenting the summarized data, individual

Protocol No. IAP312: FINAL REPORT Statistical Analysis Plan

patient response data for the efficacy analysis will be presented in Appendix 16.2. These by-patient data listings present the measurements that will be used in supporting the summary Tables. Other by-patient data listings of baseline characteristics and safety measurements will also be presented in Appendix 16.2.

# 2.14 Computer Software

All data analyses will be performed using SAS® for Windows, Release 9.1<sup>2</sup>.

#### References

- 1. Johnson, N. L. and Kotz, S. (1970), Distributions in Statistics: Continuous Univariate Distributions 1, New York: John Wiley & Sons.
- 2. SAS Release 9.1. SAS Institute Inc., Cary, North Carolina, 2004.

Table A-1 Evaluation Time Points with Evaluation Windows Used for the Summary of Global Assessment Data by Evaluation Time Point

| Evaluation<br>Time Point | Evaluation Time Point Number | Minutes from Baseline to Target Time | Evaluation Window (Minute) | | |
|---|---|---|---|---|---|
| Baseline | 0 | 1 | -14 | - | 1 |
| 2 hours | 1 | 121 | 2 | - | 181 |
| 4 hours | 2 | 241 | 182 | - | 361 |
| 8 hours | 3 | 481 | 362 | - | 721 |
| 16 hours | 4 | 961 | 722 | - | 1201 |
| 24 hours | 5 | 1441 | 1202 | - | 1681 |
| 32 hours | 6 | 1921 | 1682 | - | 2161 |
| 40 hours | 7 | 2401 | 2162 | - | 2641 |
| 48 hours | 8 | 2881 | 2642 | - | 3121 |
| 56 hours | 9 | 3361 | 3122 | - | 3601 |
| 64 hours | 10 | 3841 | 3602 | - | 4081 |
| 72 hours | 11 | 4321 | 4082 | - | 4561 |
| 80 hours | 12 | 4801 | 4562 | - | 5041 |
| Interim | X.X | | | | |

Note: Unscheduled evaluation time points and time points for premature termination are considered as regularly scheduled time points. The time point closest to the target time will be used to determine the evaluation time-specific measurement. If there are two measures that obtained at the same time distance away from the target time for the same evaluation time point number, the one prior to the target time will be used in the summary. Measures that do not fall within the evaluation windows will be considered as interim data and assigned a decimal evaluation time point number between two evaluation time point numbers in integers (e.g., 2.1 or 3.9).

Table A-2 Scheduled Evaluation Time Points with Evaluation Windows Used for the Summary of Pain Assessment Data, Blood Pressures, and Heart Rates by Evaluation Time Point

| Evaluation<br>Time Point | Evaluation Time Point Number | Minutes from Baseline to Target Time | Evaluation Window (Minute) | | |
|---|---|---|---|---|---|
| Screening | -1 | -15 | ≤ -15 | | |
| Baseline | 0 | 1 | -14 | - | 1 |
| 15 minutes | 1 | 16 | 2 | - | 23 |
| 30 minutes | 2 | 31 | 24 | - | 38 |
| 45 minutes | 3 | 46 | 39 | - | 53 |
| 1 hour | 4 | 61 | 54 | - | 91 |
| 2 hours | 5 | 121 | 92 | - | 181 |
| 4 hours | 6 | 241 | 182 | - | 301 |
| 6 hours | 7 | 361 | 302 | - | 421 |
| 8 hours | 8 | 481 | 422 | - | 541 |
| 10 hours | 9 | 601 | 542 | - | 661 |
| 12 hours | 10 | 721 | 662 | - | 841 |
| 16 hours | 11 | 961 | 842 | - | 1081 |
| 20 hours | 12 | 1201 | 1082 | - | 1321 |
| 24 hours | 13 | 1441 | 1322 | - | 1561 |
| 28 hours | 14 | 1681 | 1562 | - | 1801 |
| 32 hours | 15 | 1921 | 1802 | - | 2041 |
| 36 hours | 16 | 2161 | 2042 | - | 2281 |
| 40 hours | 17 | 2401 | 2282 | - | 2521 |
| 44 hours | 18 | 2641 | 2522 | - | 2761 |
| 48 hours | 19 | 2881 | 2762 | - | 3001 |
| 52 hours | 20 | 3121 | 3002 | - | 3241 |
| 56 hours | 21 | 3361 | 3242 | - | 3481 |
| 60 hours | 22 | 3601 | 3482 | - | 3721 |
| 64 hours | 23 | 3841 | 3722 | - | 3961 |

Protocol No. IAP312: FINAL REPORT Statistical Analysis Plan

| 68 hours | 24 | 4081 | 3962 | - | 4201 |
|----------|-----|------|------|---|------|
| 72 hours | 25 | 4321 | 4202 | - | 4441 |
| 76 hours | 26 | 4561 | 4442 | - | 4681 |
| Interim | X.X | | | | |

Note: Unscheduled evaluation time points and time points for premature termination are considered as regularly scheduled time points. The time point closest to the target time will be used to determine the evaluation time-specific measurement. If there are two measures that obtained at the same time distance away from the target time for the same evaluation time point number, the one prior to the target time will be used in the summary. Measures that do not fall within the evaluation windows will be considered as interim data and assigned a decimal evaluation time point number between two evaluation time point numbers in integers (e.g., 2.1 or 3.9).

Table A-3 Scheduled Evaluation Time Points with Evaluation Windows Used for the Summary of Respiratory Rates and Oxygen Saturation Data by Evaluation Time Point

| Evaluation<br>Time Point | Evaluation Time Point Number | Minutes from Baseline to Target Time | Evaluation Window (Minute) | | |
|---|---|---|---|---|---|
| Screening | -1 | -15 | ≤ -15 | | |
| Baseline | 0 | 1 | -14 | - | 1 |
| 15 minutes | 1 | 16 | 2 | - | 23 |
| 30 minutes | 2 | 31 | 24 | - | 38 |
| 45 minutes | 3 | 46 | 39 | - | 53 |
| 1 hour | 4 | 61 | 54 | - | 76 |
| 1.5 hours | 5 | 91 | 77 | - | 106 |
| 2 hours | 6 | 121 | 107 | - | 136 |
| 2.5 hours | 7 | 151 | 137 | - | 166 |
| 3 hours | 8 | 181 | 167 | - | 196 |
| 3.5 hours | 9 | 211 | 197 | - | 226 |
| 4 hours | 10 | 241 | 227 | - | 256 |
| 4.5 hours | 11 | 271 | 257 | - | 286 |
| 5 hours | 12 | 301 | 287 | - | 316 |
| 5.5 hours | 13 | 331 | 317 | - | 346 |
| 6 hours | 14 | 361 | 347 | - | 376 |
| 6.5 hours | 15 | 391 | 377 | - | 406 |
| 7 hours | 16 | 421 | 407 | - | 436 |
| 7.5 hours | 17 | 451 | 437 | - | 466 |
| 8 hours | 18 | 481 | 467 | - | 496 |
| 8.5 hours | 19 | 511 | 497 | - | 526 |
| 9 hours | 20 | 541 | 527 | - | 556 |
| 9.5 hours | 21 | 571 | 557 | - | 586 |
| 10 hours | 22 | 601 | 587 | - | 616 |
| 10.5 hours | 23 | 631 | 617 | - | 646 |

| 11 hours | 24 | 661 | 647 | - | 676 |
|------------|----|------|------|---|------|
| 11.5 hours | 25 | 691 | 677 | - | 706 |
| 12 hours | 26 | 721 | 707 | - | 736 |
| 12.5 hours | 27 | 751 | 737 | - | 766 |
| 13 hours | 28 | 781 | 767 | - | 796 |
| 13.5 hours | 29 | 811 | 797 | - | 826 |
| 14 hours | 30 | 841 | 827 | - | 856 |
| 14.5 hours | 31 | 871 | 857 | - | 886 |
| 15 hours | 32 | 901 | 887 | - | 916 |
| 15.5 hours | 33 | 931 | 917 | - | 946 |
| 16 hours | 34 | 961 | 947 | - | 976 |
| 16.5 hours | 35 | 991 | 977 | - | 1006 |
| 17 hours | 36 | 1021 | 1007 | - | 1036 |
| 17.5 hours | 37 | 1051 | 1037 | - | 1066 |
| 18 hours | 38 | 1081 | 1067 | - | 1096 |
| 18.5 hours | 39 | 1111 | 1097 | - | 1126 |
| 19 hours | 40 | 1141 | 1127 | - | 1156 |
| 19.5 hours | 41 | 1171 | 1157 | - | 1186 |
| 20 hours | 42 | 1201 | 1187 | - | 1216 |
| 20.5 hours | 43 | 1231 | 1217 | - | 1246 |
| 21 hours | 44 | 1261 | 1247 | - | 1276 |
| 21.5 hours | 45 | 1291 | 1277 | - | 1306 |
| 22 hours | 46 | 1321 | 1307 | - | 1336 |
| 22.5 hours | 47 | 1351 | 1337 | - | 1366 |
| 23 hours | 48 | 1381 | 1367 | - | 1396 |
| 23.5 hours | 49 | 1411 | 1397 | - | 1426 |
| 24 hours | 50 | 1441 | 1427 | - | 1501 |
| 26 hours | 51 | 1561 | 1502 | - | 1621 |
| 28 hours | 52 | 1681 | 1622 | - | 1741 |
| 30 hours | 53 | 1801 | 1742 | - | 1861 |

| 32 hours | 54 | 1921 | 1862 | - | 1981 |
|----------|-----|------|------|---|------|
| 34 hours | 55 | 2041 | 1982 | - | 2101 |
| 36 hours | 56 | 2161 | 2102 | - | 2221 |
| 38 hours | 57 | 2281 | 2222 | - | 2341 |
| 40 hours | 58 | 2401 | 2342 | - | 2461 |
| 42 hours | 59 | 2521 | 2462 | - | 2581 |
| 44 hours | 60 | 2641 | 2582 | - | 2701 |
| 46 hours | 61 | 2761 | 2702 | - | 2821 |
| 48 hours | 62 | 2881 | 2822 | - | 2941 |
| 50 hours | 63 | 3001 | 2942 | - | 3061 |
| 52 hours | 64 | 3121 | 3062 | - | 3181 |
| 54 hours | 65 | 3241 | 3182 | - | 3301 |
| 56 hours | 66 | 3361 | 3302 | - | 3421 |
| 58 hours | 67 | 3481 | 3422 | - | 3541 |
| 60 hours | 68 | 3601 | 3542 | - | 3661 |
| 62 hours | 69 | 3721 | 3662 | - | 3781 |
| 64 hours | 70 | 3841 | 3782 | - | 3901 |
| 66 hours | 71 | 3961 | 3902 | - | 4021 |
| 68 hours | 72 | 4081 | 4022 | - | 4141 |
| 70 hours | 73 | 4201 | 4142 | - | 4261 |
| 72 hours | 74 | 4321 | 4262 | - | 4441 |
| 76 hours | 75 | 4561 | 4442 | - | 4681 |
| Interim | X.X | | | | |

Note: Unscheduled evaluation time points and time points for premature termination are considered as regularly scheduled time points. The time point closest to the target time will be used to determine the evaluation time-specific measurement. If there are two measures that obtained at the same time distance away from the target time for the same evaluation time point number, the one prior to the target time will be used in the summary. Measures that do not fall within the evaluation windows will be considered as interim data and assigned a decimal evaluation time point number between two evaluation time point numbers in integers (e.g., 2.1 or 3.9).